CLINICAL TRIAL: NCT00318734
Title: Trace Elements and CVD Risk Factors Among Young Adults
Brief Title: Examining the Link Between Trace Elements and Cardiovascular Disease Risk Factors in Young Adults
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1335; R01HL081572-01A1 (NIH)
Record Dates: First submitted 2006-04-25; First posted 2006-04-27 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2011-12

CONDITIONS: Cardiovascular Diseases; Metabolic Syndrome X; Hypertension; Inflammation; Atherosclerosis
MeSH Terms: conditions — Cardiovascular Diseases; Metabolic Syndrome; Hypertension; Inflammation; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Cardiovascular disease (CVD) affects millions of people in the United States; each year, more people die from CVD than from any other disease. There are many dietary and lifestyle factors that may increase the risk of developing CVD. Preliminary research has shown that the presence of certain trace elements may be associated with the development of CVD. This study will examine toenail clippings and laboratory data to evaluate the link between trace elements and CVD risk factors in young adults.

DETAILED DESCRIPTION:
CVD is a disorder that affects the heart's ability to function normally. The most common cause of heart disease is narrowing or blockage of the coronary arteries, which supply blood to the heart. There are many risk factors for CVD, including inflammation, high blood pressure, high cholesterol, and obesity. Small quantities of trace elements, also known as micronutrients, are essential in maintaining a healthy body. Research has shown that some trace elements may be associated with the development of CVD, but more research is needed to confirm this connection. This study will examine concentrations of several trace elements in toenail samples of young adults participating in the Coronary Artery Risk Development in Young Adults (CARDIA) study. The CARDIA study is measuring changes in CVD risk factors in individuals as they age and is identifying lifestyle habits that influence those changes. The purpose of this study is to determine the link between trace elements and CVD risk factors in young adults. The results of this study may help to identify whether dietary, lifestyle, or environmental factors can be modified at a young age to prevent the development of CVD.

This study will examine laboratory and medical history data of participants who are already enrolled in the CARDIA study; there are no additional study visits specifically for this study. Toenail samples collected from participants during their Year 2 CARDIA study visit in the late 1980's will be examined to determine the presence of selenium, chromium, arsenic, and mercury. Participants' CARDIA study data will be reviewed and several CVD risk factors will be analyzed, including the thickness of heart arteries; calcium buildup within the arteries; inflammatory markers, such as high sensitivity C-reactive protein and interleukin 6; blood pressure levels; body weight; and levels of cholesterol, fat, and sugar.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the CARDIA study; this current study will be using existing CARDIA study data and will not be recruiting any new participants

Ages: 20 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participating in the CARDIA study.
Sampling Method: Non-Probability Sample
Enrollment: 4362 (Actual)
Dates: Start 2006-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
CVD risk factors | 1987-2010

CONTACTS AND LOCATIONS:
Overall Officials: Ka He, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States